CLINICAL TRIAL: NCT06305819
Title: Managing Symptoms and Disability in the Sub-acute Phase After Traumatic Injury - A Pragmatic Randomised Controlled Trial of a Self-management Support Program
Brief Title: Effectiveness of a Self-management Program After Traumatic Injury
Acronym: SEMPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Sunnaas Rehabilitation Hospital (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Nada Andelic, Head of Research and Development, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023057
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Trauma Injury; Trauma, Multiple; Polytrauma
Keywords: Self-management program; Rehabilitation; Sub-acute phase
MeSH Terms: conditions — Accidental Injuries; Multiple Trauma | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants assigned to intervention arm will receive the self-management support program. The program consists of 2.5-hour sessions and is delivered to groups of 5-7 participants. The intervention is provided over a period of eight weeks with one session per week and is delivered by a multidisciplinary team. A tele-health version of the intervention will be offered to those who prefer to participate via electronic devices.
  Interventions: Behavioral: self-management support program
- Control (Active Comparator): Participants assigned to the control group will receive the usual health and rehabilitation services provided in the municipality or other rehabilitation settings. These services will potentially vary greatly from no services to specialized or local rehabilitation teams. All services received by participants in the control group will be registered at the follow-ups.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: self-management support program — The SEMPO program is inspired by established self-management principles and established rehabilitation strategies. The program is manualized and integrates components from rehabilitation strategies within relevant functional domains. The program includes elements, such as tailored psychoeducational content, action planning, guided skills mastery, learning and practicing helpful compensatory strategies, problem solving techniques and sharing of experiences. The intervention is delivered by a multidisciplinary team and the participants are provided with written materials and a work book containing information about each session and work tasks.
  Other Names: SEMPO
  Arms: Intervention
Other: Control group — Treatment as usual
  Other Names: Control
  Arms: Control

SUMMARY:
Traumatic injuries, defined as a physical injury with sudden onset, are a leading cause to disability and impaired health. Persons who sustain a traumatic injury often report problems in daily life activities and reduced quality of life, which may limit participation in work/studies, leisure activities and family life. Consequently, complex rehabilitation and support is recommended in National Trauma guidelines due to the often long-lasting physical and psychological sequela of the injury.

The main goal of this study is to determine the effectiveness of a self-management support program delivered to persons with a moderate or severe traumatic injury in the sub-acute phase of recovery (i.e. 3-4 months after injury). The self-management program aims to enhance patients' self-efficacy by building skills and self-management strategies to cope with injury-related consequences. The program has a group-based format and consists of eight sessions comprising psychoeducation, skill mastery and sharing of experiences. The participants who will be included in the study must be between 18 and 70 years, be residing in the southeast region of Norway, be admitted to Oslo University hospital or transferred from local hospital within 72 hours after injury, have at least a two-day hospital stay, and be able to read and understand Norwegian language. Participants will be randomly assigned to either intervention or control group. A group of patients will also be able to self-select if they want to receive the self-management support program or be in the control group. The latter is an explorative part of the study to evaluate the influence of patients' treatment-preferences on the study outcomes. Participants in the control group will receive treatment as usual.

DETAILED DESCRIPTION:
This study is designed as a pragmatic randomized controlled trial using a mixed-methods design with 6-months follow-up to determine the effectiveness of a newly developed self-management support program, entitled the SEMPO. Participants will be included 3-4 months post-injury and followed up over a 12 months period.

Study setting and participants:

The study will be conducted at Oslo University Hospital (OUH). Patients will be recruited at the Trauma Centre at Oslo University Hospital, which is the Level 1 trauma centre for the southeast region of Norway and serves a population base consisting of more than half of the Norwegian population. Patients who fulfil the following inclusion criteria will be asked to participate:

* Adults residing in the southeast region of Norway who are aged between 18 and 72 years.
* Admitted to OUH directly or after transfer from local hospitals within 72 hours of injury.
* At least a two-day hospital stay.
* Traumatic injury corresponding to a New Injury Severity Scale score (NISS) >9.
* Patients reporting injury-related symptoms, functional impairments, and/or difficulties with daily activities at the discharge from OUH. According to preliminary analyses in ongoing study on unmet needs after trauma (funded by South-Eastern Norway Regional Health Authority), these patients are in risk of developing long-lasting disabilities.

Patients will be excluded in case of:

* Cognitive function corresponding to a Mini Mental Status score (MMS) < 20 points.
* Psychiatric diseases that require treatment.
* Drug/alcohol dependence that require treatment.
* Complete spinal cord injury and isolated thoracic or abdominal injury.
* Insufficient command of Norwegian.

Patients who consent to participate will be randomised into a randomisation arm (RA) or a self-selection arm (SA). Participants in the RA will then be further randomised to intervention or control group. In the self-selection arm, the participants can choose whether they will be placed in the intervention or control group. The self-selection arm is an explorative part of the study to explore if taking into account patient treatment preferences may maximise adherence, reduce potential attrition bias and influence the intervention results. Data will be collected through interview/patient-reported outcome measures (PROMs) at the following time points: baseline assessment (T1), after completion of the intervention (T2), 3-months after completion of the intervention (T3), and 6-months after the intervention (T4), with similar time-points for those in the control group.

The primary outcome is self-efficacy assessed with the Trauma Coping Self-Efficacy Scale. Secondary outcomes include symptom burden, physical, cognitive and emotional functioning. Additional outcomes include resilience, health-related quality of life, communication with health professionals, health literacy, global functioning and disability, and evaluation of changes. The participants will complete all outcome measures. In addition, participants will nominate their target problem areas with their own words and will be asked to select one personal outcome preference from the predefined outcomes.

Sample size calculation and statistical analyses:

Sample size was estimated based on the primary outcome. Results from a study on mental eHealth interventions following trauma were used. A power calculation was conducted with a standard deviation of 1.0 and a mean group difference of 0.6. Given an 80% power and an alpha of 0.05, 90 participants should be included to observe significant treatment related improvement. With an assumed attrition rate of 20%, 110 participants will be included (i.e. 55 participants in each group). The sample size calculation was done based on the randomization arm (RA), and we aim to achieve the same power in the self-selection (SA) arm. However, the SA is considered an exploratory part of this study to evaluate the influence of patients' treatment preferences.

To investigate the effectiveness of the intervention on self-efficacy, symptom burden and disability, and patient-impression of change, mixed-effect models will be used to account for repeated measurements by patients. Time and time-by-treatment interaction will be used as fixed effects in these models. The linear mixed model will give estimated mean values for all time points (T1, T2, T3, and T4), changes from baseline, and between -group differences from baseline with 95% confidence intervals. The analyses will be based on an "intention to treat" principle. In addition, clinical benefit will be estimated in quality-adjusted life years (QALYs) using standardized conversion tools to convert health benefits into an index of HRQL, as measured by EQ-5D. Simulated cost consequences of the program will be considered from health and societal perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Adults residing in the southeast region of Norway who are aged between 18 and 72 years.
* Admitted to OUH directly or after transfer from local hospitals within 72 hours of injury.
* At least a two-day hospital stay.
* Traumatic injury corresponding to a New Injury Severity Scale score (NISS) >9.
* Patients reporting injury-related symptoms, functional impairments, and/or difficulties with daily activities at the discharge from OUH.

Exclusion Criteria:

* Cognitive function corresponding to a Mini Mental Status score (MMS) < 20 points.
* Psychiatric diseases that require treatment.
* Drug/alcohol dependence that require treatment.
* Complete spinal cord injury and isolated thoracic or abdominal injury
* Insufficient command of Norwegian

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Trauma Coping Self-Efficacy | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in self-efficacy in trauma coping, measured on a 9-item questionnaire, with Likert scale from 1 (not capable) to 7 (totally capable).

SECONDARY OUTCOMES:
Rivermead Post-Concussion Symptom Questionnaire | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in post-concussion symptoms measured on a 16-item questionnaire, with Likert scale from 0 (no symptoms) to 4 (severe symptom)
Fatigue Severity Scale | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in fatigue symptoms measured on a 9-item questionnaire, with a Likert scale from 1 (Totally disagree) to 7 (totally agree).
Insomnia Severity Index | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in sleep disturbance measured on a 5-item questionnaire, with Likert scale from 1-5.
Brief Pain Inventory -short form | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in pain measured on a 9-item questionnaire, with Likert scale from 0 -10.
International Physical Activity Questionnaire | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported frequency of physical activity and specific levels of intensity.
Cognitive Failures Questionnaire | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in cognitive failures measured on a 25-item questionnaire, with Likert scale from 0 (never) to 4 (very often).
Patient Health Questionnaire-9 | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in depressive symptoms measured on a 9-item questionnaire, with Likert scale from 0 (not at all) to 3 (nearly every day).
Generalised Anxiety Disorder-7 | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in anxiety symptoms measured on a 7-item questionnaire, with Likert scale from 0 (not at all) to 3 (nearly every day).
Impact of Event Scale - Revised | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in post-traumatic stress symptoms measured on a 22-item questionnaire, with Likert scale from 0 (not at all) to 4 (extremely).
Return to work | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-report of full-time/part-time job (percentage); hours per week

OTHER OUTCOMES:
Resilience Scale for Adults | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in post-traumatic stress symptoms measured on a 33-item questionnaire, with Likert scale from 0 to 4.
EuroQol five-dimensional questionnaire | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-reported change in health-related quality of life measured on a 5-item questionnaire, with Likert scale from 1 to 5.
Target Outcomes | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Self-nominated 3 most troublesome difficulties related to trauma injury. Problem area rated how difficult it is to manage the problem on a five-point Likert scale from 0 (not at all difficult) to 4 (extremely difficult).
Patient Global Impression of Change | Change immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  One- item questionnaire measuring self-evaluation in global change of functioning, on a Likert scale from 1 (no change) to 7 (a great deal better).
Intervention acceptability and satisfaction | Measured immediately after the intervention period (T2).
  Intervention group only. 8-item questionnaire measuring level of satisfaction and program
  usefulness on a Likert scale from 1 (not useful) to 5 (extremely useful).
Intervention satisfaction | Measured immediately after the intervention period (T2).
  Intervention group only. Open-ended questionnaire inquiring satisfaction with intervention.
WHO Disability Assessment Scale | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  12-item questionnaire measuring health and disability on a Likert scale from 1 (no difficulty) to 5 (extremely difficult).
Glasgow Outcome Scale - Extended | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  The GOS-E is an ordinal scale measuring global functioning outcome: (1) Death, (2) Vegetative State, (3) Lower Severe Disability, (4) Upper Severe Disability, (5) Lower Moderate Disability, (6) Upper Moderate Disability, (7) Lower Good Recovery, and (8) Upper Good Recovery.
Communication with physicians | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  3-item questionnaire measuring degree of coping in communication with health care providers, measured on a Likert scale from 0 (never) to 5 (always)
Health Literacy Questionnaire | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  3-item questionnaire measuring level of health literacy, measured on a Likert scale from 1 (always a problem) to 5 (never)
Received health care services | Change from baseline (T1) to immediately after the intervention period (T2), 3 months after intervention (T3), and 6 months after intervention (T4)
  Type and frequency of health care services received

CONTACTS AND LOCATIONS:
Overall Officials: Nada Andelic, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Only aggregated data will be shared according to the Norwegian legislation

REFERENCES:
- [Derived] Rasmussen MS, Andelic N, Selj JN, Danielsen VM, Lovstad M, Howe EI, Hellstrom T, Soberg HL, Brunborg C, Aas E, Moksnes H, Sveen U, Gaarder C, Naess PA, Helseth E, Roise O, Aarhus M, Ora HP, Bjorneboe JA, Fure S, Roe C, Schafer C, Perrin PB, Lu J, Elf M, Dahl HM, Jones F, Ponsford J, Narvestad L, Hauger SL. Self-management support program delivered in the sub-acute phase after traumatic injury-study protocol for a pragmatic randomized controlled trial. Trials. 2024 Sep 30;25(1):639. doi: 10.1186/s13063-024-08492-0. PMID 39350137